CLINICAL TRIAL: NCT06408142
Title: Universal Test and Connect for HIV Service Delivery in South Africa and Baltimore
Brief Title: Universal Test and Connect for HIV Service Delivery in South Africa
Acronym: UTC: SA
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Desmond Tutu HIV Foundation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00443103; 1R34MH138250 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Human Immunodeficiency Virus; Pre-Exposure Prophylaxis; Emergency Department; South Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Emergencies | interventions — HIV Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency Department Patients in South Africa: Universal Test and Connect: universal screening with HIV testing followed by demographic/clinical information to determine number of patients who would be eligible for HIV PrEP
  Interventions: Diagnostic Test: HIV testing
- Emergency Department Providers: Nurses, physicians, or advanced practice providers who deliver care in the Emergency Department at one of the clinical sites
  Interventions: Other: In-depth interview

INTERVENTIONS:
Diagnostic Test: HIV testing — Point of Care HIV testing universally regardless of risk factors
  Groups: Emergency Department Patients in South Africa
Other: In-depth interview — In-depth interviews of providers using Normalization Process Theory semi-structured interview guide to assess provider perspectives of PrEP delivery in the ED
  Groups: Emergency Department Providers

SUMMARY:
The goal of this study is to determine how many patients with HIV or at high risk of getting HIV attend the Emergency Department (ED) in South Africa (SA). The investigators will integrate HIV assessment in the ED and see how many people who would be a candidate for a drug that prevents HIV (PrEP). Universal test and connect (UTC) is a strategy that universally tests all patients and connects patients to long-term care, whether HIV positive or negative, including referrals for PrEP. The investigator's goal is to use UTC across two busy 24-hr EDs in Cape Town, SA.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to deliver comprehensive HIV services for patients with HIV or at high risk of HIV acquisition attending the Emergency Department (ED) in South Africa (SA). The investigators seek to integrate HIV assessment in the ED and define the opportunity for delivering biomedical HIV prevention interventions in this setting. EDs provide care to high volumes of adults who may not otherwise interact with the health system, and thus are an important testing and linkage to care venue. Access to both preventative (pre- and post-exposure prophylaxis) and therapeutic (ART (antiretroviral) initiation) HIV services from the ED can expand care to otherwise missed populations and aligns directly with a differentiated service delivery model that is integrated within existing, sustainable service delivery models.

Universal test and connect (UTC) is a holistic strategy that endeavors to accelerate the race to reduce new HIV infections and deaths from AIDS-related illnesses. Trials in Africa have shown that within three years of implementing a community-wide UTC program, HIV incidence decreased by 20-30%, and AIDS-related mortality decreased by 20% . This strategy resulted in increased diagnosis among men and provided preventative resources to young women. Given ED patients' vulnerabilities and lack of access to routine services, UTC is a new and needed tool to provide comprehensive ED-based HIV services. Currently, testing is haphazard, and while occupational exposure may be addressed, preventative strategies for other high-risk exposures are not.

The investigators seek to demonstrate that the ED has a high volume of patients that could potentially benefit from HIV services (i.e., HIV testing, ART initiation, pre-exposure prophylaxis (PrEP)/post-exposure prophylaxis (PEP) initiation, and linkage to care) and that HIV service delivery in this venue is necessary and feasible to integrate. Furthermore, the investigators seek to explore the missed opportunity to deliver PrEP in the ED, thus expanding PrEP access to all segments of the population. The investigators propose to demonstrate that PrEP initiation in the ED is an important investment to providing holistic care for ED patients and that providers will be accepting of ED-based PrEP delivery if HIV testing and PrEP initiation can be effectively integrated into clinical workflow.

ELIGIBILITY:
Inclusion Criteria for universal testing and connecting:

* Patients attending the Emergency Department
* Ages > or = 12 years old in South Africa
* For subset that participate in PrEP choice trial, inclusion criteria will be to ensure that they meet PrEP eligibility criteria and do not have any contraindications to PrEP (kidney disease, acute HIV signs or symptoms, already taking PrEP).

Exclusion Criteria:

* Patients unable to provide written informed consent - i.e., have a depressed level of consciousness (head trauma or concurrent alcohol/substance abuse), determined as critically ill (triage score of "emergent"), or
* do not speak a language spoken by the study team (English, Afrikaans, and Xhosa).

In-depth interviews and surveys to providers:

Inclusion Criteria:

* Nurses, physicians, or advanced practice providers (APPs) who work regularly in the Emergency Department at one of the clinical sites.
* Consent to a recorded in-depth interview and/or Normalizing Process Theory (NPT) survey

Exclusion Criteria:

* Providers who have already been interviewed (if working at both clinical sites)
* Providers who do not consent to an interview or a survey.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cross-sectional population attending the Emergency Departments, which are both publicly available 24-hour Emergency Departments that serve the surrounding neighborhood/catchment area.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of potentially PrEP eligible patients in the ED | Baseline
  Baseline survey, chart abstraction, and use of South Africa National Department of Health and Centers for Disease Control and Prevention (CDC) pre-exposure prophylaxis (PrEP) Eligibility Guidelines

SECONDARY OUTCOMES:
The number of potentially PrEP eligible patients with tuberculosis or acute HIV | Baseline
  Lab testing obtained through medical record
The number of potentially PrEP eligible patients with renal dysfunction | Baseline
  Lab testing obtained through medical record
The number of potentially PrEP eligible patients who report baseline difficulty to engage in follow up required to be on PrEP | Baseline
  Social Determinants of Health Survey including financial insecurity (1-5), food insecurity (two questions, one 1-4 and the other 1-5), transportation needs (yes vs no as need for transportation within past 12 months), physical activity level (days per week of exercise and average exercise time per exercise session), stress (1-5), social connections (1-5), substance use (number of drinks or use off illicit substances used per week), intimate partner violence (Number of instances in past 12 months). Scored on subscales, parentheses indicating Likert scores with lower scores indicating worse outcome
Acceptability of ED PrEP to ED Providers | after implementation of UTC

CONTACTS AND LOCATIONS:
Overall Officials: Bhakti Hansoti, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Gugulethu Community Health Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers that are explicitly on the IRB (Institutional Review Board) both at Johns Hopkins or on local IRBs at University of Cape Town and Stellenbosch University. All information will be de-identified while not on an encrypted password-protected database to ensure participant confidentiality
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Throughout duration of study period (anticipated 2027) and up to 5 years after.
Access Criteria: Researchers/analysts on the Institutional Review Board (IRB) submission at each of the IRB sites for this multi-center study